CLINICAL TRIAL: NCT01210313
Title: Physical Activity for Reduction of Recurrence Rate After Adjuvant Chemotherapy for Localised Colorectal Carcinoma
Status: Completed | Type: Observational
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: ABCSG C07; EXERCISE (Other: ABCSG)
Record Dates: First submitted 2010-09-23; First posted 2010-09-28 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Carcinoma
Keywords: physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical exercise: No treatment, only physical examinations accompanying physical exercise
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Defined exercise program

SUMMARY:
* feasibility of physical activity
* increase of physical conversation
* Quality of Life (optional)
* vascular and metabolic effects

DETAILED DESCRIPTION:
In this phase II pilot project the feasibility of a defined medical physical activity should be verified for increased physical conversation. The study is conducted multicentric (single group) with a study population of 30 patients. After completion of adjuvant chemotherapy the patients will participate a defined physical training, 3 times per week within a time period of 52 weeks. Planned study duration 2 years.

ELIGIBILITY:
Inclusion Criteria:

* complete resected, histologically confirmed adeno carcinoma of colon or rectal and condition after (neo-)adjuvant therapy either in (1) stage III or (2) stage II with risk factor
* 4-16 weeks after the end of an adjuvant chemotherapy
* ECOG 0,1
* Age > 18 years
* adequate liver-, nephro- and hemogram parameters
* physical eligibility

Exclusion Criteria:

* significant comorbidities which exclude the participation
* evidence of local recurrence or distant metastases
* non-compliance of subject
* other malignancy within the last 5 years (except: skin basalioma, cervix carcinoma in situ)
* clinically significant cardiovascular diseases
* treatment with beta blocker without possibility of adjustment
* left bundle-branch block
* simultaneous chemotherapy or radiotherapy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with localised colorectal carcinoma
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Thaler, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group; Michael Fridrik, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group; Alfred Fridrik, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (7):
- Austria (7):
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - Medical University Innsbruck, Internal Medicine, Innsbruck, Tyrol
  - District Hospital Kufstein, Kufstein, Tyrol
  - AKH Linz, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - State Hospital Rankweil, Rankweil, Vorarlberg
  - Paracelsus Medical University Salzburg-Oncology, Coop. Group, Salzburg

REFERENCES:
- [Result] Meyerhardt JA, Giovannucci EL, Holmes MD, Chan AT, Chan JA, Colditz GA, Fuchs CS. Physical activity and survival after colorectal cancer diagnosis. J Clin Oncol. 2006 Aug 1;24(22):3527-34. doi: 10.1200/JCO.2006.06.0855. Epub 2006 Jul 5. PMID 16822844
- [Result] Meyerhardt JA, Heseltine D, Niedzwiecki D, Hollis D, Saltz LB, Mayer RJ, Thomas J, Nelson H, Whittom R, Hantel A, Schilsky RL, Fuchs CS. Impact of physical activity on cancer recurrence and survival in patients with stage III colon cancer: findings from CALGB 89803. J Clin Oncol. 2006 Aug 1;24(22):3535-41. doi: 10.1200/JCO.2006.06.0863. Epub 2006 Jul 5. PMID 16822843
- [Result] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Result] Demark-Wahnefried W. Cancer survival: time to get moving? Data accumulate suggesting a link between physical activity and cancer survival. J Clin Oncol. 2006 Aug 1;24(22):3517-8. doi: 10.1200/JCO.2006.06.6548. Epub 2006 Jul 5. No abstract available. PMID 16822842
- [Result] Jackson AS, Pollock ML. Generalized equations for predicting body density of men. Br J Nutr. 1978 Nov;40(3):497-504. doi: 10.1079/bjn19780152. PMID 718832
- [Result] Hoeger W, Hoeger S. Principles and Labs for Physical Fitness. Morton Publishing Company, first edition 1999
- [Result] O'Donovan G, Owen A, Bird SR, Kearney EM, Nevill AM, Jones DW, Woolf-May K. Changes in cardiorespiratory fitness and coronary heart disease risk factors following 24 wk of moderate- or high-intensity exercise of equal energy cost. J Appl Physiol (1985). 2005 May;98(5):1619-25. doi: 10.1152/japplphysiol.01310.2004. Epub 2005 Jan 7. PMID 15640382
- [Result] Haber Paul. Leitfaden zur medizinischen Trainingsberatung - Rehabilitation bis Leistungssport. 3. Auflage 2009; Springer Wien New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled October 7, 2010, the last participant was enrolled March 22, 2012. Enrollment took place in 7 Austrian clinical sites. In total, 30 participants were enrolled.
Groups:
- Physical Exercise: No treatment, only physical examinations accompanying physical exercise (defined exercise program)
Period: Overall Study
Arm/Group | Physical Exercise
Started | 30
Completed | 14
Not Completed | 16
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Distant recurrence | 4
Not completed — Non-compliance | 7

BASELINE CHARACTERISTICS:
Population: One among the 30 enrolled participants had both colon and rectum cancer and only information from rectum cancer is given in the baseline.
Groups:
- Total: All participants (patients with colorectal cancer after adjuvant chemotherapy) included in this single arm study.
Arm/Group | Total
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Cancer location [Count of Participants; unit: Participants]
  Colon | 12
  Rectum | 17
  Colon and rectum | 1
pT-Stage [Count of Participants; unit: Participants] — Pathologic T-stage: pT1, tumour only in the inner layer of the bowel; pT2, tumour has grown into the muscle layer of the bowel wall; pT3, tumour has grown into the outer lining of the bowel wall but has not grown through; pTX, not determinable
  Participants
    pT1 | 4
    pT2 | 4
    pT3 | 16
    pT4 | 5
    pTX | 1
pN-Stage [Count of Participants; unit: Participants] — Pathologic N-stage: pN0, no lymph nodes containing cancer cells; pN1, cancer cells in 1 to 3 nearby lymph nodes or in the nearby tissue; pN2, cancer cells in 4 or more nearby lymph nodes
  Participants
    pN0 | 10
    pN1 | 14
    pN2 | 6
Chemotherapy [Count of Participants; unit: Participants]
  Adjuvant | 19
  Adjuvant and neoadjuvant | 11
Height [Median (Full Range); unit: cm] | 175 [160 to 192]
Weight [Median (Full Range); unit: kg] | 76 [51 to 134]
pM-Stage [Count of Participants; unit: Participants] — Pathologic M-stage (metastases): M0, the cancer has not spread to other organs; MX: not determinable
  Participants
    pM0 | 27
    pMX | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Physical Activity After 12 Weeks (3 Months)
Description: Evaluation of the feasibility measured in terms of training adherence during the first 12 weeks measured in actual participant-weeks in relation to the 360 planned participant-weeks during cycle 1 (week 1 to week 12)
Time Frame: 3 months
Population: Total of all 30 participants enrolled
Measure: Count of Units; unit: Participant-weeks
Units Other Than Participants: Participant-weeks
Arm/Group | Physical Exercise
Number analyzed (Participants) | 30
Number analyzed (Participant-weeks) | 360
Participant-weeks | 331

2. Primary Outcome: Feasibility of Physical Activity After 26 Weeks (6 Months)
Description: Evaluation of the feasibility measured in terms of training adherence during the weeks 13 to 26 measured in actual participant-weeks in relation to the planned 420 participant-weeks during cycle 2 (week 13 to week 26)
Time Frame: 6 months
Population: Total of all 30 participants enrolled
Measure: Count of Units; unit: Participant-weeks
Units Other Than Participants: Participant-weeks
Arm/Group | Physical Exercise
Number analyzed (Participants) | 30
Number analyzed (Participant-weeks) | 420
Participant-weeks | 277

3. Primary Outcome: Feasibility of Physical Activity After 52 Weeks (12 Months)
Description: Evaluation of the feasibility measured in terms of training adherence during the weeks 27 to 52 measured in actual participant-weeks in relation to the planned 780 participant-weeks during cycle 3 (week 27 to week 52)
Time Frame: 12 months
Population: Total of all 30 participants enrolled
Measure: Count of Units; unit: Participant-weeks
Units Other Than Participants: Participant-weeks
Arm/Group | Physical Exercise
Number analyzed (Participants) | 30
Number analyzed (Participant-weeks) | 780
Participant-weeks | 468

4. Secondary Outcome: Exercise Ergometry Activity After 12 Weeks (3 Months)
Description: Evaluation by exercise ergometry and descriptively compared with the planned exercise ergometry after 12 weeks; measured in mean METs (metabolic equivalent of task) per week in relation to the planned mean 10 METs during cycle 1 (week 1 to week 12)
Time Frame: 3 months
Population: All participants with METs information
Measure: Mean (Standard Deviation); unit: kcal/kg/hour
Arm/Group | Physical Exercise
Number analyzed (Participants) | 21
kcal/kg/hour | 9.43 (7.82)

5. Secondary Outcome: Exercise Ergometry Activity After 26 Weeks (6 Months)
Description: Evaluation by exercise ergometry and descriptively compared with the planned exercise ergometry after 26 weeks; measured in mean METs (metabolic equivalent of task) per week in relation to the planned mean 15 METs during cycle 2 (week 13 to week 26)
Time Frame: 6 months
Population: All participants with METs information
Measure: Mean (Standard Deviation); unit: kcal/kg/hour
Arm/Group | Physical Exercise
Number analyzed (Participants) | 18
kcal/kg/hour | 12.7 (7.23)

6. Secondary Outcome: Exercise Ergometry Activity After 52 Weeks (12 Months)
Description: Evaluation by exercise ergometry and descriptively compared with the planned exercise ergometry after 52 weeks; measured in mean METs (metabolic equivalent of task) per week in relation to the planned mean 18 METs during cycle 3 (week 27 to week 52)
Time Frame: 12 months
Population: All participants with METs information
Measure: Mean (Standard Deviation); unit: kcal/kg/hour
Arm/Group | Physical Exercise
Number analyzed (Participants) | 14
kcal/kg/hour | 11.27 (8.61)

7. Secondary Outcome: Adiponectin at Screening
Description: Evaluation of adiponectin at screening as baseline for a description of changes during the study
Time Frame: Day 1 (at screening)
Population: All participants with information on adiponectin
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 20
μg/ml | 9.93 (2.88)

8. Secondary Outcome: Adiponectin After 12 Weeks (3 Months)
Description: Evaluation of adiponectin after 12 weeks (3 months) for a description of changes during the study
Time Frame: 3 months
Population: All participants with information on adiponectin
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 19
μg/ml | 8.14 (3.79)

9. Secondary Outcome: Adiponectin After 52 Weeks (12 Months)
Description: Evaluation of adiponectin after 52 weeks (12 months) for a description of changes during the study
Time Frame: 12 months
Population: All participants with information on adiponectin
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 14
μg/ml | 9.31 (3.37)

10. Secondary Outcome: Leptin at Screening
Description: Evaluation of leptin at screening as baseline for a description of changes during the study
Time Frame: Day 1 (at screening)
Population: All participants with information on leptin
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 20
ng/ml | 36.02 (31.68)

11. Secondary Outcome: Leptin After 12 Weeks (3 Months)
Description: Evaluation of leptin after 12 weeks (3 months) for a description of changes during the study
Time Frame: 3 months
Population: All participants with information on leptin
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 19
ng/ml | 41.12 (43.07)

12. Secondary Outcome: Leptin After 52 Weeks (12 Months)
Description: Evaluation of leptin after 52 weeks (12 months) for a description of changes during the study
Time Frame: 12 months
Population: All participants with information on leptin
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Physical Exercise
Number analyzed (Participants) | 14
ng/ml | 42.5 (41.74)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Physical Exercise
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Exercise (N=30)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Heart pain (Cardiac disorders) | 1 (2)
Indisposition (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No